CLINICAL TRIAL: NCT05516277
Title: Insomnia Treatment and Cardiometabolic Health in Older Adults With Posttraumatic Stress Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Monica R. Kelly, PhD, DBSM, Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1K23HL157754-01A1 (NIH)
Record Dates: First submitted 2022-08-16; First posted 2022-08-25 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Posttraumatic Stress Disorder; Insomnia; Cardiovascular Diseases; Metabolic Disease
Keywords: Quality of Life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Cardiovascular Diseases; Metabolic Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: All eligible participants will receive the same treatments for PTSD and insomnia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Sleep Education Intervention (Experimental): Manual-based education program focusing on behavioral sleep techniques provided in individual 60-minute sessions for 5 weekly sessions.
  Interventions: Behavioral: Behavioral Sleep Education Intervention

INTERVENTIONS:
Behavioral: Behavioral Sleep Education Intervention — Manual-based education program focusing on behavioral sleep techniques provided in individual 60-minute sessions for 5 weekly sessions.
  Other Names: Cognitive Behavioral Therapy for Insomnia

SUMMARY:
This pilot pre-post trial will address a gap in knowledge related to addressing modifiable risk factors for cardiometabolic disease through treating residual insomnia, sleep difficulties that remain after successful treatment of another condition, in the context of PTSD in understudied older adults. This study provides a non-medication treatment for PTSD called Cognitive Processing Therapy (CPT) followed by a non-medication sleep education and treatment program (Cognitive Behavioral Therapy for Insomnia, CBT-I) for sleep problems that remain after completing PTSD treatment in older adults with PTSD. The aims of this project are to evaluate 1) the added benefits of treating residual insomnia on sleep and PTSD symptoms; 2) the added benefits of treating residual insomnia following CPT on cardiometabolic risk biomarkers and quality of life; and 3) the durability of the sleep, PTSD, cardiometabolic and quality of life benefits of treating residual insomnia following CPT at 6-month follow-up in older adults with PTSD.

DETAILED DESCRIPTION:
Both insomnia and Post Traumatic Stress Disorder (PTSD) are independent risk factors for cardiometabolic diseases; the leading causes of morbidity and mortality in the US for which the growing geriatric population is at elevated risk. PTSD and insomnia disorder frequently co-occur yet require unique treatments, as sleep difficulties are one of the most common residual symptoms that remain after completing an evidence-based PTSD treatment.

This pilot pre-post trial provides a non-medication treatment for PTSD called Cognitive Processing Therapy (CPT) followed by a non-medication sleep education and treatment program (Cognitive Behavioral Therapy for Insomnia, CBT-I) for sleep problems that remain after completing PTSD treatment in older adults with PTSD. Individuals over 50 years of age, who have received care at the VA Greater Los Angeles Healthcare System, and who have been exposed to a stressful or traumatic life event will be recruited for this study.

Participants will be asked to complete a baseline evaluation that involves (a) being asked questions about health, medications, personal information, quality of life, sleep patterns and habits, mood, and stressful/traumatic experiences; (b) wearing a blood pressure monitor at home for 24 hours; (c) wearing a continuous glucose monitor sensor that contains a small filament (a thread-sized needle) inserted into the upper arm or abdomen for 7 consecutive days; (d) wearing a wristwatch device that measures sleep/wake patterns for 7 consecutive days; and (e) completing a daily sleep diary for 7 consecutive days. Participants may also be screened for sleep apnea with a portable sleep apnea monitoring device with sensors worn on the wrist, index finger and chest for one night.

Information from the baseline evaluation and medical records will be reviewed by the research team to determine whether an individual is eligible and likely able to complete all future study activities. Participants will be contacted to be advised of their study eligibility status. If eligible after the baseline assessment, study staff will review future study activities and confirm the participant's interest in continuing in the study. All eligible and interested participants will then receive an evidence-based PTSD treatment (CPT; 12 sessions). Following completion of the PTSD treatment, participants will receive a sleep education program (CBT-I; 5 sessions). For eligible individuals, participation in this research will last about 11 months.

Main study outcomes assessments from the baseline evaluation will be repeated three times: (1) one week after completion of the PTSD treatment; (2) one week after completion of the sleep education program; and (3) 6-months after the sleep education program ends. Data will be analyzed using "intention to treat" principles, using appropriate statistical methods for pilot clinical trials.

The investigators hope to determine how these treatment programs affect health in older adults with PTSD and insomnia. Findings from this pilot study will expand our understanding of the relationships between evidence-based insomnia and trauma treatments and key outcomes of sleep, PTSD symptoms, cardiometabolic health and quality of life in older adults with PTSD and insomnia while informing future research.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling Veterans aged 50 years and older
* Received care from a Veterans Health Administration (VHA) facility in the prior year
* Diagnosis of PTSD
* Diagnosis of insomnia disorder
* Lives within a 50-mile radius of the research offices at the VA Sepulveda Ambulatory Care Center

Exclusion Criteria:

* Active substance use or in recovery with less than 90 days of sobriety
* Too ill to engage in the study procedures (e.g., unable to attend the in-person meetings)
* Unable to self-consent to participate
* Unstable housing (as this will impact the research team's ability to retrieve costly and difficult to replace monitoring equipment)
* Severe cardiovascular or respiratory disease (e.g., ventilatory failure, CHF)
* Unstable medical or psychiatric disorders (which are a contraindication for behavioral treatment of insomnia)
* Comorbid sleep disorders (i.e., central sleep apnea syndrome, diagnosed narcolepsy or circadian rhythm sleep-wake phase disorders) based on medical record review and baseline assessment data, or untreated, severe sleep disordered breathing (SDB) as assessed via WatchPAT or previous clinical evaluation (apnea-hypopnea index [AHI] ≥ 30; or AHI ≥ 15 plus Epworth Sleepiness Scale [ESS] score ≥ 10) that better explain sleep difficulties

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Consensus sleep diary questionnaire | Change from baseline to 1 week after completion of sleep intervention
  Self-reported sleep quality assessed with the Consensus sleep diary, a brief patient questionnaire evaluating multiple aspects of sleep quality including sleep onset latency (time to fall asleep in minutes) and sleep efficiency percentage (time asleep in minutes/time in bed in minutes x 100).
PTSD Checklist for DSM-5 (PCL-5) | Change from baseline to 1 week after completion of sleep intervention
  The PCL-5 is a self-report PTSD severity questionnaire evaluating multiple aspects of PTSD symptoms. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. A higher score indicates more severe PTSD symptoms.
24-hr ambulatory blood pressure monitoring (ABPM) blood pressure variability | Change from baseline to 1 week after completion of sleep intervention
  ABPM is an assessment of hypertension, a cardiometabolic disease, and blood pressure patterns across the 24-hour period. We will assess within-subject blood pressure variability via standard deviation across 24-hours.
24-hr ambulatory blood pressure monitoring (ABPM) systolic/diastolic loads | Change from baseline to 1 week after completion of sleep intervention
  ABPM is an assessment of hypertension, a cardiometabolic disease, and blood pressure patterns across the 24-hour period. We will assess systolic/diastolic loads via percentage of elevated values across 24-hours.
24-hr ambulatory blood pressure monitoring (ABPM) change in blood pressure day to night | Change from baseline to 1 week after completion of sleep intervention
  ABPM is an assessment of hypertension, a cardiometabolic disease, and blood pressure patterns across the 24-hour period. We will assess change in blood pressure from day to night (day-night).
WHOQOL-BREF questionnaire | Change from baseline to 1 week after completion of sleep intervention
  Self-reported quality of life assessed with a brief patient questionnaire evaluating aspects of quality of life across four domains: 1) Physical health, 2) Psychological, 3) Social relations, and 4) Environment. Mean scores for each domain range from 4-20, which are multiplied by 4 to transform the domain score into a scaled score that is comparable to the full WHOQOL-100 measure. A higher score indicated higher quality of life.

SECONDARY OUTCOMES:
Homeostatic Model Assessment of Insulin Resistance (HOMA) | Change from baseline to 1 week after completion of sleep intervention
  HOMA is an assessment of insulin resistance, a cardiometabolic disease risk factor
Hemoglobin A1c (HbA1c) | Change from baseline to 6 months after completion of sleep intervention
  HbA1c is an assessment of hyperglycemia, a cardiometabolic disease.
Body Mass Index (BMI) | Change from baseline to 1 week after completion of sleep intervention
  BMI is a measure body composition, a cardiometabolic disease risk factor.
Central adiposity | Change from baseline to 1 week after completion of sleep intervention
  Hip-to-waist ratio is a measure of central adiposity, a cardiometabolic disease risk factor.
Actigraphy | Change from baseline to 1 week after completion of sleep intervention
  Actigraphy is a wrist-watch style device with an imbedded accelerometer that measures movement to define sleep/wake patterns including sleep onset latency (time to fall asleep) and sleep efficiency (time asleep/time in bed x 100).
Dyslipidemia | Change from baseline to 1 week after completion of sleep intervention
  Fasting serum lipids are measures of dyslipidemia, a cardiometabolic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Kelly, PhD, Principal Investigator — UCLA / VA Greater Los Angeles
Locations (1):
- VA Greater Los Angeles Healthcare System, North Hills, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data (IPD) available to other researchers as this is a pilot study.

DOCUMENTS (1):
  • Informed Consent Form (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT05516277/ICF_002.pdf